CLINICAL TRIAL: NCT03482037
Title: Effects of Two Different Doses of Rec 0/0438 Administered by Intravesical Instillation in Patients With Neurogenic Detrusor Overactivity Due to Spinal Cord Injury: a Repeated Doses, Double-blind, Placebo Controlled Study
Brief Title: Effects of Rec 0/0438 in Patients With Neurogenic Detrusor Overactivity Due to Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Rec 0/0438-IT-CL 0491; 2017-000905-19 (EudraCT Number)
Record Dates: First submitted 2018-03-08; First posted 2018-03-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Neurogenic Detrusor Overactivity

STUDY DESIGN:
Intervention Model Description: two sequential cohorts, each corresponding to a dose level.
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rec 0/0438 (Experimental): Rec 0/0438 1 mg (first cohort), 2 mg (second cohort) to be administered by intravesical instillation once daily for four weeks
  Interventions: Drug: Rec 0/0438 1 mg or Rec 0/0438 2 mg
- Placebo (Placebo Comparator): Placebo, to be administered by intravesical instillation once daily for four weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rec 0/0438 1 mg or Rec 0/0438 2 mg — Each vial content will be administered via the catheter used for the self-catheterization
  Arms: Rec 0/0438
Drug: placebo — Each vial content will be administered via the catheter used for the self-catheterization
  Arms: Placebo

SUMMARY:
Study to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of Rec 0/0438 in subjects with neurogenic detrusor overactivity due to spinal cord injury

DETAILED DESCRIPTION:
Multicentre, double-blind, randomised, parallel groups, placebo-controlled study to be conducted in specialized centres in Europe to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of two different doses of Rec 0/0438 in comparison with placebo, in subjects with neurogenic detrusor overactivity due to spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥18 years and ≤65 years.
* Female subjects must be either sterile or, if with child-bearing potential, must have a pregnancy test negative and commit to the use of a highly effective method of birth control (see Appendix 15.6) for the duration of the study, and until at least 1 month after the last dose of study medication. Male subjects must be willing to use male contraception (condom) to avoid pregnancies of their female partner of childbearing potential throughout the entire duration of the study, and for 3 months after the last dose of study medication.
* Suffering from NDO due to SCI at upper motor neuron level (below C6) and emptying the bladder performing clear intermittent self-catheterization (CISC).
* Subjects classified in group A, B, or C, of the ASIA (American Spinal Injury Association) impairment scale.
* Stable therapy for NDO in the last thirty days (Subjects should maintain the therapy stable for the duration of the study).
* At least 1 incontinence episode/day despite current treatment, according to what is reported in the Bladder Diary filled in by the subject.
* Subjects with diastolic blood pressure values between 60 and 99 mmHg (both inclusive), and systolic blood pressure values between 90 and 159 mmHg (both inclusive). Blood pressure measurement must be performed in subjects with an empty bladder.
* Subjects with stable concomitant medication treatment at baseline.
* Written informed consent must be given by subjects before any study related investigational procedures is performed.

Exclusion Criteria:

* Breastfeeding women.
* Treatment with injection of botulinum toxin, unless in the opinion of the Investigator the bladder activity has returned to pre-treatment level.
* Use of prohibited concomitant medications, such as drugs that could affect immunoassay testing (systemic corticosteroids: prednisone, budesonide, prednisolone; calcineurin inhibitors: cyclosporine, tacrolimus; mTOR inhibitors: sirolimus, everolimus; IMDH inhibitors: azathioprine, leflunomide, mycophenolate; biologics: abatacept, adalimumab, anakinra , certolizumab, etanercept, golimumab, infliximab, ixekizumab, natalizumab, rituximab, secukinumab, tocilizumab, ustekinumab, vedolizumab; monoclonal antibodies: basiliximab, daclizumab, muromonab) or initiation of therapy with drugs affecting lower urinary tract symptoms (such as alpha-blockers, tadalafil 5 mg oad). If already present at Screening visit, therapy with drugs affecting lower urinary tract symptoms must be maintained stable through the study period (Note: occasional treatment with PDE-5 inhibitors for erectile dysfunction should be avoided between Screening visit and Day 8 and between Day 25 and 28).
* History of cerebro- or cardio-vascular diseases (TIA, stroke, hypertensive encephalopathy, angina pectoris, MI, cardiac by-pass, CHF NYHA classes III and IV).
* Uncontrolled type 1 or type 2 diabetes (Hb A1c >8 %).
* Moderate to severe renal impairment (estimated creatinine clearance <60 mL/min by the Cockcroft-Gault equation).
* Moderate to severe liver impairment (any liver function test: AST, ALT, GGT, Bilirubin >2.5 times the upper limit of normal).
* Hemodynamically significant valve disease, including aortic stenosis or clinically significant ventricular or supraventricular arrhythmia, heart rate >100 beats/min.
* Clinically important abnormal laboratory findings during the run-in period, including: Haemoglobin <10 g/dL; Serum Potassium >5.5 mmol/L; Serum Sodium <132 mmol/L.
* Symptomatic active urinary tract infection (i.e. cloudy and/or malodorous urine, chills, fever, increased muscle spasticity or increased autonomic dysreflexia, letargy, hypotension, malaise).
* Evidence of any neoplastic disease.
* History of allergy, hypersensitivity or intolerance to drugs.
* Participation in an investigational drug study within 30 days prior to the screening assessment.
* Any other diseases or conditions, that according to the Investigator's opinion, make the subject unable to comply with protocol requirements, or unable to complete the study or increases the risk to the subject or which prevents optimal participation in achieving the objectives of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Day 28
  Treatment-emergent adverse events occurred with treatment with Rec 0/0438

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | Day 1 and Day 7
  Peak Plasma Concentration (Cmax)
Area Under the Curve (AUC) | Day 1 and Day 7
  Area under the plasma concentration versus time curve (AUC)
Change from baseline in Maximum Cystometric Capacity | Day 28
  The volume at which uncontrollable voiding begins during filling Cystometry

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Cruz, M.D., Principal Investigator — Hospital São João, Urologia, Alameda Prof. Hernâni Monteiro, 4200-319 Porto, Portugal
Locations (9):
- Recordati Investigative Site, Prague, Czechia
- France (4):
  - Department of Urology, Academic hospital Pitié-Salpêtrière, Assistance Publique-Hôpitaux de Paris, Pierre et Marie Curie Medical School, Sorbonne Universités, Paris
  - Centre Hospitalier Lyon Sud Unité de Pharmacie Clinique Oncologique (essai clinique) Pavillon Marcel Bérard - Bât. 1G, Pierre-Bénite
  - Recordati Investigative Site, Rouen
  - Recordati Investigative Site, Toulouse
- Poland (3):
  - Recordati Investigative Site, Piaseczno
  - Recordati Investigative Site, Rzeszów
  - Recordati Investigative Site, Warsaw
- Recordati Investigative Site, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No